CLINICAL TRIAL: NCT05020483
Title: Activated Prothrombin Complex Concentrate FEIBA to Optimize Postcardiopulomonary Bypass Hemostasis in Pediatric Cardiac Patients
Brief Title: FEIBA to Optimize Postcardiopulmonary Bypass Hemostasis in Pediatric Cardiac Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Patient population changed and no subjects eligible for the study.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Elena Ashikhmina, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-005539
Record Dates: First submitted 2021-08-18; First posted 2021-08-25 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Cardiac Disease
Keywords: Cardiac Surgery
MeSH Terms: conditions — Heart Diseases | interventions — anti-inhibitor coagulant complex

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FEIBA Group (Experimental): Pediatric patients ≤15 kg of weight, undergoing cardiac surgery with cardiopulmonary bypass will receive activated prothrombin complex concentrate (aPCC) FEIBA to be incorporated into standard treatment of post-bypass coagulopathic bleeding.
  Interventions: Drug: FEIBA
- Placebo Group (Placebo Comparator): Pediatric patients ≤15 kg of weight, undergoing cardiac surgery with cardiopulmonary bypass will receive a placebo to be incorporated into standard treatment of post-bypass coagulopathic bleeding.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FEIBA — Administered via the central line catheter after termination of cardiopulmonary bypass if bleeding related to poor clotting develops; in addition, according to conventional protocol blood products will be transfused simultaneously. Three small doses, 5 mg/kg each, will be available.
  Other Names: activated prothrombin complex concentrate (aPCC) FEIBA
  Arms: FEIBA Group
Drug: Placebo — Contains no active ingredient and administered via the central line catheter after termination of cardiopulmonary bypass if bleeding related to poor clotting develops; in addition, according to conventional protocol blood products will be transfused simultaneously.
  Arms: Placebo Group

SUMMARY:
The purpose of this research is to understand if the medication called FEIBA helps to stop bleeding and decrease transfusion of blood products to small children operated on the heart.

ELIGIBILITY:
Inclusion Criteria:

* Weight ≤ 15 kg.
* Elective cardiac surgery with cardiopulmonary bypass.
* Coagulopathic bleeding after cardiopulmonary bypass.
* Availability and willingness of the parent/legal guardian to provide informed consent.

Exclusion Criteria:

* Presence of mechanical circulatory support at the time of randomization or POD 0 and 1.
* Patient or family history of coagulopathy and/or thromboses.
* Preoperative anticoagulation (excluding low dose heparin for "line prophylaxis").

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of units of allogeneic blood products required early perioperatively in pediatric cardiac patients. | approximately 1 day postoperatively
  Number of units of transfused allogeneic blood products after cardiopulmonary bypass in the operating room (OR) and in the intensive care unit (ICU) on postoperative day (POD) 0 and 1.

SECONDARY OUTCOMES:
Hospital length of stay | Through hospital discharge, approximately 3 days
  Number of days admitted to the hospital
Mortality | Through hospital discharge, approximately 3 days
  Total number of subject deaths
Intravascular and intracardiac thromboses | approximately 3 days postoperatively
  Number of subjects to experience intravascular and/or intracardiac thromboses up to POD 3

CONTACTS AND LOCATIONS:
Overall Officials: Elena Ashikhmina, MD, PhD, Principal Investigator — Mayo Clinic

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials